CLINICAL TRIAL: NCT04053933
Title: A Multicenter Observational Belgian Study Assessing the Impact of Newly Started Treatment on the QOL in Patients Suffering From Myelodysplastic Syndromes.
Brief Title: Observational Study Towards the Impact of Newly Started Treatment in MDS on QoL
Acronym: Be-QUALMS
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Zwi Berneman, Professor, University Hospital, Antwerp
Other Study IDs: B300201938708
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Myelodysplastic Syndromes
Keywords: QUALMS; MDS; Be-QUALMS; Quality of life; QoL
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Patients treated with ESA
- Patients treated with 5'azacitidin
- Patients treated with deferoxamine
- Patients treated with deferasirox
- Patients treated with transfusion only
- Patients treated with lenalidomide
- Patients treated with intensive chemotherapy

SUMMARY:
Study type An observational study conducted in different hematological centers in Belgium.

Study objectives

Primary objective:

To assess the impact of newly started treatments on the QOL of patients suffering from myelodysplastic syndromes.

Secondary objectives:

* To assess the impact of newly started therapy on disease perception in MDS patients
* To study the relation between disease perception and quality of life
* To examine which clinical and disease specific factors determine QOL in MDS patients
* Collect information on the transfusion threshold in Belgian hematological centers and evaluate the impact on quality of life.
* To evaluate whether changes in QOL are related to hematological respons.

Study design

* Newly diagnosed MDS patients who are about to start a treatment or previously diagnosed MDS patients who are starting with a new line of therapy.
* QOL assessment with the QUALMS.
* Disease perception measurement using the B-IPQ.
* Measurement at diagnosis/before start of therapy, at 4 weeks, 12 weeks, and at 24 weeks into treatment.

Study endpoints

Primary endpoint:

Change in QUALMS score at visit timepoints 4 - 12 - 24 weeks after the start of a new treatment.

Secondary endpoint:

* Change in B-IPQ score at visit timepoints 4 - 12 - 24 weeks after the start of a new treatment
* Association between B-IPQ and QUALMS score.
* Association between clinical and disease specific factors and QUALMS score
* Association between transfusion threshold and QUALMS score.
* Association between hematological response and QUALMS score

Summary of eligibility criteria

* Adult patients with a new diagnosis of MDS (according to WHO 2016 definitions (3) or known patients with MDS who are about to start a new treatment.
* Signed informed consent.
* Patients enrolled in an unblinded interventional therapeutic trial are eligible.

Exclusion criteria

* Patients with acute leukemia defined as >20% bone marrow blasts.
* Patients suffering from an overlap syndrome myelodysplastic/myeloproliferative disease.
* Patients in post allogeneic transplant setting.
* Patients enrolled in a blinded interventional therapeutic trial.
* Patients starting with multiple treatments under investigation at the same moment apart from intensive chemotherapy.
* Newly diagnosed patients who do not start with treatment.
* Patients who started a previous treatment less then 12 weeks ago apart from packed cell transfusion (up to 4 weeks allowed).
* Diagnosis of any previous or concomitant malignancy except when the patient successfully completed treatment (chemotherapy and/or surgery and/or radiotherapy) with curative intent for this malignancy at least 3 months prior to inclusion.
* Patients refusing to sign informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with myelodysplastic syndromes defined by WHO 2016 criteria that are about to start treatment.
* Patients with a known diagnosis of MDS, irrespective of IPSS and irrespective of time of diagnosis that are about to start a new therapy.
* Signed informed consent

Exclusion criteria

* Patients with acute leukemia defined as >20% bone marrow blasts.
* Patients suffering from a myelodysplastic/myeloproliferative overlap syndrome. In this case the disease has both dysplastic and proliferative features but cannot be properly categorized to either group. This category includes chronic myelomonocytic leukemia (CMML), juvenile myelomonocytic leukemia (JMML), atypial chronic myeloid leukemia (aCML) and myelodysplastic/myeloproliferative disease unclassifiable.
* Patients in post allogeneic transplant setting.
* Patients enrolled in a blinded interventional therapeutic trial.
* Patients starting with multiple MDS treatments at the same moment apart from intensive chemotherapy.
* Newly diagnosed patients who do not start with treatment.
* Patients who started a previous MDS related treatment less then 4 weeks ago.
* Patients who started a previous MDS related treatment less then 12 weeks ago apart from packed cell transfusions.
* Diagnosis of any previous or concomitant malignancy except when the patient successfully completed treatment (chemotherapy and/or surgery and/or radiotherapy) with curative intent for this malignancy at least 3 months prior to inclusion.
* Patients refusing to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from myelodysplastic syndromes
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in QUALMS-score | 6 months
  Change in quality of life-score after the start of a new MDS related treatment
Change in IPQ-score | 6 months
  Change of ilness perception score after the start of a new MDS related treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zwi Berneman, MD,PhD, Principal Investigator — University Hospital, Antwerp
Locations (21):
- Belgium (21):
  - Imelda, Bonheiden, Antwerpen
  - AZ KLINA, Brasschaat, Antwerpen
  - Sint-Dimpna Ziekenhuis Geel, Geel, Antwerpen
  - Heilig Hart Ziekenhuis, Lier, Antwerpen
  - UZA, Edegem, Antwerp
  - CH Jolimont, La Louvière, Henegouwen
  - CHR Mons Hainaut, Mons, Henegouwen
  - CHU Ambroise Paré, Mons, Henegouwen
  - CHU - UCL Namur site Godinne, Yvoir, Namur
  - UZ Gent, Ghent, Oost Vlaanderen
  - AZ Nikolaas, Sint-Niklaas, Oost Vlaanderen
  - Institute Jules Bordet, Brussels, Vlaams Brabant
  - UZ Brussel, Jette, Vlaams Brabant
  - UZ Leuven Gasthuisberg, Leuven, Vlaams Brabant
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert, Vlaams Brabant
  - AZ Sint Jan Brugge, Bruges, West Vlaanderen
  - AZ Damiaan Oostende, Ostend, West Vlaanderen
  - Ziekenhuis Netwerk Antwerpen, Antwerp
  - GasthuisZusters Antwerpen, Antwerp
  - CHR Namur, Namur
  - BR Clinic Saint Pierre Ottignies, Ottignies-Louvain-la-Neuve

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heyrman B, Meers S, De Becker A, Wouters K, Van Hoof A, Van De Velde A, Graux C, Mazure D, Selleslag D, Maes H, Lemmens J, Beckers M, Breems D, Sid S, Berneman Z, Anguille S. Disease Perception Is Correlated with Health-Related Quality of Life in Patients Suffering from Myelodysplastic Syndromes: Results of the Belgian Be-QUALMS Study. Cancers (Basel). 2023 Jun 22;15(13):3296. doi: 10.3390/cancers15133296. PMID 37444406

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT04053933/Prot_SAP_000.pdf